CLINICAL TRIAL: NCT06936228
Title: Evaluation of the Effect of Local Propolis Application on the Healing of Pressure Sores
Brief Title: Evaluation of the Effect of Local Propolis Application on the Healing of Pressure Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Cigdem Kuralay, Lecturer, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Çiğdem Kuralay; Çiğdem KURALAY (Registry Identifier: Propolis Application in Pressure Ulcer")
Record Dates: First submitted 2025-03-24; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Pressure Sore
Keywords: Pressure ulcer; Propolis application; Apitherapy
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 Propolis (Experimental): Propolis was applied in addition to standard wound treatment administered in the hospital for 21 days.
  Interventions: Dietary Supplement: Propolis spray
- 2 control (No Intervention): The control group received standard wound care treatment administered in the hospital for 21 days, and the researcher did not intervene in any way.

INTERVENTIONS:
Dietary Supplement: Propolis spray — The product obtained from 30% pure Anatolian propolis was applied once daily.
  Arms: 1 Propolis

SUMMARY:
The study was conducted to evaluate the effect of local propolis application in patients with pressure ulcers. A total of 62 patients were included in this randomized controlled experimental study, with 31 patients in the propolis group and 31 in the control group. While the control group received the clinic's standard wound care treatment protocol, the propolis group was administered 30% pure propolis extract in addition to the standard wound care treatment protocol. For data collection, the following tools were used: the Introductory Characteristics Form, which includes patients' socio-demographic and medical information; the Propolis Application Follow-up Form; the Pressure Ulcer Healing Assessment Scale; pain assessment tools including the Visual Analog Scale (VAS) for conscious patients and the Face Pain Scale for unconscious patients; Katz's Index of Activities of Daily Living; and the Charlson Comorbidity Index (CCI).

ELIGIBILITY:
Inclusion Criteria:

The patient or their caregiver is able to communicate verbally, Hospitalized in palliative care or intensive care units for at least one week, Has a Stage 1, 2, or 3 pressure ulcer according to NPUAP (13), The wound has not been closed by a physician, Agrees to participate in the study, Expected to stay in the hospital for at least 21 days.

Exclusion Criteria:

The patient or their caregiver is unable to communicate verbally, Has a Stage 4 or unstageable pressure ulcer according to NPUAP, The wound has been closed by a physician, Does not agree to participate in the study, Expected to stay in the hospital for less than 21 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Pressure Ulcer Healing: PUSH (Pressure Ulcer Scale for Healing) | 21-day follow-up
  It was developed by the EPUAP (European Pressure Ulcer Advisory Panel) to monitor changes in pressure ulcers. It includes three subdimensions: tissue type, exudate amount, and pressure ulcer area. To calculate the pressure ulcer area, the length and width of the wound are multiplied, resulting in a value in cm². This value is then evaluated on a 10-point scale. The amount of exudate is scored as follows: none - 0 points, slight - 1 point, moderate - 2 points, and heavy - 3 points. The third subdimension, tissue type, is scored as follows: 4 points if there is necrotic tissue, 3 points if there is no necrotic tissue but eschar is present, 2 points if granulation tissue is present and the wound is clean, 1 point if epithelialization is observed, and 0 points if the wound is completely closed. The total score, ranging from 0 to 17, provides information about the condition of the ulcer. An increase in the score indicates greater severity of the ulcer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bakanlığı Ordu Üniversitesi Eğitim ve Araştırma Hastanei, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No